CLINICAL TRIAL: NCT06222437
Title: Semaglutide and Polycystic Ovarian Syndrome: an Emerging Treatment Strategy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 046.OBG.2023.D
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Protocol group (Experimental): PCOS women in the age 18 to 45 years
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — effectiveness of semaglutide in PCOS

SUMMARY:
The purpose of this study is to investigate the effect of semaglutide in women with Polycystic Ovarian Syndrome(PCOS ) and determine potential therapeutic benefits.

DETAILED DESCRIPTION:
The study mainly focused for the following objectives:

To determine the effect of semaglutide on ovulation and menstrual regularity. To determine the effect of semaglutide on androgen levels, namely testosterone, sex hormone binding globulin, and changes in hirsutism.

To determine changes in weight, body mass index (BMI), and Glycated Hemoglobin( HbA1c) with semaglutide therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Body mass index(BMI) > 30
* Diagnosis of PCOS
* Normal thyroid stimulating hormone, prolactin, follicle-stimulating hormone (FSH), estradiol, and normal progesterone

Exclusion Criteria:

* Medications excluded: any hormone-containing contraceptive - oral contraceptive pills, Progesterone-only pill, depo-provera, oral provera, progesterone-containing intrauterine contraceptive device
* Letrozole, clomiphene citrate, FSH therapy
* Androgen receptor blockers
* 5α reductase inhibitors
* Insulin
* Hysterectomy
* Endometrial ablation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with PCOS
Enrollment: 85 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of appropriate weekly dose | 4 weeks
  To access the compliances of the therapy
Number of days on therapy | 4 weeks
  To access the persistence on Semaglutide

SECONDARY OUTCOMES:
measure the Weight in kilograms | 4 weeks
  To access the weight changes during therapy
Numbers of days with exercise changes | 4 weeks
  To access the ability to do exercise during the therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Institute at Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No